CLINICAL TRIAL: NCT02715323
Title: Exploring Immune Cell Signatures in Autoimmunity and Ocular Surface Stress
Brief Title: Exploring Immune Cell Signatures in Autoimmunity and Dry Eye Syndrome
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: SingHealth Translational Immunology and Inflammation Centre (Unknown); TTSH Eye Clinic (Unknown)
Responsible Party: Principal Investigator, Louis Tong, Principal Investigator, Singapore National Eye Centre
Other Study IDs: R1295/101/2015 (SERI-STIIC-3); 2016/2048 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Autoimmunity; Dry Eye Syndrome
Keywords: dry eye; immunological profile; autoimmune
MeSH Terms: conditions — Autoimmune Diseases; Dry Eye Syndromes | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cross-sectional study

SUMMARY:
Ocular surface disease, especially dry eye and scleritis, commonly affects patients with autoimmune diseases. Ocular surface immune cells are increased in autoimmune disease; however the full subset of immune cells activated is unknown. Recent experimental studies show that dendritic cells and T cells in the cornea are critically associated with corneal nerve innervation. Corneal confocal microscopy (CCM) allows rapid non-invasive in vivo imaging of dendritic cells and corneal nerves. The investigators propose to investigate how ocular surface health, conjunctival immune cells and corneal nerve/dendritic cell morphology interact in 3 rheumatological conditions: Sjogren's syndrome (SS), Rheumatoid arthritis (RA), Systemic lupus erythematosus (SLE).

The preliminary flow cytometric studies show that various immune cells (eg: T cells, B cells, and dendritic cells) can be quantified using minimally invasive impression membranes (Eyeprim). Clinically, the research team is experienced in measuring features of ocular surface inflammation (conjunctival redness, tear breakup times) with Oculus keratograph5M. The investigators also aim to harvest conjunctival immune cells using impression cytology and quantify specific cell types with flow cytometry. Corneal nerve morphology and dendritic cell density and distribution will be assessed using CCM; in collaboration with the group who have pioneered this technique.

The investigator anticipate that alterations in corneal nerve and dendritic cell parameters will correlate with immune activation/inflammation, deterioration of tear function and increased systemic severity of the rheumatological disease. In addition, the investigators hypothesize that the lower the corneal nerve density, the higher the number of corneal dendritic cells and conjunctival inflammatory cells. Studying these relationships may allow a better mechanistic understanding of local corneal and systemic immune activation and the development of a non-invasive ophthalmic surrogate marker of dendritic cell activation and nerve fibre loss to aid earlier diagnosis, risk stratification and the development of new therapies in autoimmune patients with severe dry eye.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE

   1.1 General Introduction

   Ocular surface disease, especially dry eye and scleritis, commonly affects patients with autoimmune diseases. Ocular surface immune cells are increased in autoimmune disease; however the full subset of immune cells activated is unknown. Recent experimental studies show that dendritic cells and T cells in the cornea are critically associated with corneal nerve innervation. Corneal confocal microscopy (CCM) allows rapid non-invasive in vivo imaging of dendritic cells and corneal nerves. The investigators propose to investigate how ocular surface health, conjunctival immune cells and corneal nerve/dendritic cell morphology interact in 3 rheumatological conditions: Sjogren's syndrome (SS), Rheumatoid arthritis (RA), Systemic lupus erythematosus (SLE).

   The preliminary flow cytometric studies show that various immune cells (eg: T cells, B cells, and dendritic cells) can be quantified using minimally invasive impression membranes (Eyeprim). Clinically, the research team is experienced in measuring features of ocular surface inflammation (conjunctival redness, tear breakup times) with Oculus keratograph5M. The investigators also aim to harvest conjunctival immune cells using impression cytology and quantify specific cell types with flow cytometry. Corneal nerve morphology and dendritic cell density and distribution will be assessed using CCM; in collaboration with the group who have pioneered this technique.

   Investigators anticipate that alterations in corneal nerve and dendritic cell parameters will correlate with immune activation/inflammation, deterioration of tear function and increased systemic severity of the rheumatological disease. In addition, the investigator hypothesize that the lower the corneal nerve density, the higher the number of corneal dendritic cells and conjunctival inflammatory cells. Studying these relationships may allow a better mechanistic understanding of local corneal and systemic immune activation and the development of a non-invasive ophthalmic surrogate marker of dendritic cell activation and nerve fibre loss to aid earlier diagnosis, risk stratification and the development of new therapies in our autoimmune patients with severe dry eye.

   1.2 Rational for the Study Purpose

   Dry eye, a type of chronic ocular surface inflammation, is highly prevalent and contributes to corneal blindness and imposes a severe health burden. Scleritis is ocular surface inflammatory disorder associated with mild to severe inflammation of the sclera with or without intraocular inflammation. Severe dry eye or scleritis is associated with autoimmune diseases like SS, RA, SLE, and other conditions. Current treatment of dry eye is often not effective enough (eg., cyclosporine) or causes adverse effects (eg., corticosteroid-induced glaucoma). In autoimmune dry eye, there is immune-mediated damage to the ocular surface and the lacrimal gland. In various models of dry eye disease, it has been shown that components of the immune system such as T cells, macrophages and cytokines such as interleukin (IL) 1β and tumor necrosis factor (TNF)-α are critical for triggering and maintaining this disease. Likewise treatment of non-infective sclerits is a very challenging situation to all uveitis specialists.

   Ocular surface immune cells are increased when autoimmune disease is present, either the proportion or number of a particular type of immune cell, eg. monocytes or CD4+ T cells may be increased in the presence of more severe local inflammation and/or systemic activity. A signature of immune cell infiltration may be present in a particular rheumatological condition. If certain types of cells, (e.g., T cells or B cells) are predominant in the systemic disease, it suggests that a T cell approach (e.g., tacrolimus) or B cell approach (e.g., rituxamab) may be used. Alternatively, if certain cytokines play a major role in dry eye, an inhibitor of cytokine signalling such as a JAK inhibitor may be used.

   Recent studies have shown that dendritic cells and T cells in the cornea are critically associated with corneal nerve innervation [1, 2]. This has been shown in both human and animal studies [1-4]. At the same time, the technology for in vivo imaging of human corneal nerves and dendritic cells and their quantification have greatly improved recently. This has led to an explosion of interest in harnessing this technology as a surrogate marker for peripheral neuropathies and to explore underlying mechanisms [5-27]. The investigators have previously shown that first generation CCM can quantify the presence and density of Langerhans cells (LCs) in Bowman's layer of the cornea in patients with diabetes [28]. However the latest 3rd generation HRT III can be used to classify and quantify Langerhans cells (LCs) into a mature phenotype (dendritic cell bearing long processes) or an immature phenotype (non-dendritic cell lacking cell dendrites) to provide insight into immune alterations in vivo [29]. A recent experimental study in diabetic mice has used CCM to show that direct contact between DCs and the corneal nerves may trigger nerve fiber damage [30].

   Gap in scientific knowledge: Researchers have shown that proinflammatory cytokines are elevated in tears of humans with dry eye; many of these may be secreted by immune cells. They found in preliminary flow cytometric studies that CD4+ T cells, CD19+ B cells, CD14+ monocytes, CD1c dendritic cells can be quantified using minimally invasive impression membranes (Eyeprim)[31]. The full subset of immune cells activated in the ocular surface in dry eye, and in various rheumatological conditions, is not known. The proportions of these cells in different severity of dry eye and different systemic activity of autoimmune disease have not been evaluated. Furthermore, it is uncertain whether the integrity of cornea innervation is also a determinant of tear function in patients with autoimmune systemic disease.

   The research group has undertaken many clinical trials and imaging studies of the human ocular surface. This includes measurements with Oculus (non-invasive tear breakup times), staining, etc., and the measurement of cytokines using the multiplex bead based sandwich immunofluorescence assay[32-38]

   Preliminary Studies The research group has also optimized Eyeprim collection of conjunctival immune cells and method of analysis using a panel of immune markers with Amnis [31], a relatively new type of flow cytometry (Figure 1) coupled with microscopy (Figure 2). The advantage of the Amnis technique is the direct visualization of analyzed cells to permit co-localisation of signals. They have published on the validity of the cell morphological parameter analysis using the Amnis software, compared to a human grader [31]. In addition, they have also used conventional flow cytometry (BD FACS) to quantify CD3, CD4, CD8, CCR7, CXCR3, CD109 and CD63 staining (data not shown).

   In collaboration with the ENA team, their team has been trained in image acquisition using CCM to enable quantification of corneal nerves and dendritic cells [1, 2, 4, 9, 10, 13, 14, 16, 21, 27](Figure 3). Sub-basal corneal nerve fibre density, corneal nerve branch density, corneal nerve fibre length and tortuosity (Figure 3, 4) will be quantified using both manual (CCMetrics) and automated (ACCMetrics) image analysis software, developed by the ENA team. Sub-basal mature and immature dendritic cell density and distribution in relation to corneal nerves will be quantified.

   The collaborators, Prof Malik and Dr. Petropoulos are leading the Early neuropathy assessment (ENA team-http://qatar-weill.cornell.edu/research/faculty/eng/index.html) and have pioneered the use of in vivo CCM as a rapid, non-invasive ophthalmic instrument to monitor diabetic and other peripheral neuropathies. They will actively engage in training and overseeing optimal image capture and will provide the necessary software and licensing privileges to enable detailed quantification and interpretation [9, 10, 12-14, 16, 17, 20, 21, 23-27].
2. HYPOTHESIS AND OBJECTIVES Overall long term objective: Discover safe and effective treatment for ocular surface inflammation and define the ocular surface indications for clinical usage of medications targeting the immune system in rheumatological disease.

   Clinical / Healthcare implications: There are many benefits in using CCM in autoimmune disease. CCM allows rapid, non-invasive imaging of the corneal nerves and dendritic cells to determine the level of inflammation and its consequence in autoimmune diseases. This will allow earlier diagnosis, risk stratification and more timely intervention at the rheumatology clinics, enhancing multidisciplinary care of autoimmune patients. The investigator will build a normative database (either ethnic or local age specific data from a reading centre) by using this study as a platform to recruit more patients.

   Basic science implications: Advance understanding of relationship between corneal nerves and tear function/immunology.

   Short term objectives: researchers propose a nationwide study in collaboration with Tan Tock Seng Hospital to study clinical features and conjunctival immune cells in patients with ocular surface inflammatory disease with or without associated systemic autoimmune or collagen vascular disease.

   Academic objectives: Aim to:
   * Enhance multidisciplinary collaborations, between SERI and S Albani from STIIC (cell analysis)
   * Build new collaborations (TTSH ophthalmologist Dr R Agrawal)
   * Increase value/synergy from currently approved funding: SERI pilot grant (recruitment of pilot participants and optimization of tools),
   * Compete for future funding, NMRC STAR award, CS or CBIRG.

   Expected findings:
   * Different systemic severities of the rheumatological diseases, symptoms of dry eye, tear function, NIKBUT and corneal staining may correlate with corneal nerve and dendritic/non-dendritic cell defects.
   * Tear cytokines may correlate with corneal nerve and dendritic/non-dendritic cell defects.
   * Change in the density and subtypes of T cells or other cells such as dendritic in the conjunctiva (impression cytology) may correlate with corneal nerve and dendritic/non-dendritic cell defects.

   2.3 Potential Risks and Benefits: 2.3.1 Potential Risks
   * It is possible that there may be some slight discomfort during the sampling of conjunctival cells using the impression membrane
   * Some slight discomfort or redness from tear fluid collection (Schirmer test)
   * Rarely a corneal epithelial defect may occur from in vivo confocal microscopy, but this generally heals in 1-2 days. Corneal epithelial defect means that a layer of the cornea is broken, liken to what happened during an abrasion.
   * Stinging sensation as a result of local anaesthetic (Alcaine)

   2.3.2 Potential Benefits With greater understanding of the presence of various inflammatory mediators, the investigators can gain further insight into the complex process taking place in autoimmune diseases patients.
3. STUDY POPULATION 3.1 List The Number and Nature of Subjects to be Enrolled. The investigators will recruit patients with 3 specific rheumatological diagnoses and controls

   * SS (n=40), RA (n=40), SLE (n=40)
   * Healthy age/ethnicity/sex matched control subjects (n=40)

   Total sample size: 160
4. STUDY DESIGN This is a cross-sectional study involving 160 participants. Study duration: One visit, recruitment duration: 1 Year

4.1.1 Screening Visit and Procedures Screening visit and procedures will be done on a separate day. Participants referred from TTSH will be allocated a time slot to come to SERI for the ocular examinations. On the day of procedure, SERI coordinator will screen for eligible subjects by asking them some questions base on the inclusion and exclusion checklist. If found to be eligible and participants are interested, consent will be taken at SERI and SERI optometrist will proceed with the ocular assessments.

4.1.2 Study Procedures

The examinations will be done by SERI study team members. The list of required examinations is shown:

1. Dry Eye Symptoms (SPEED Questionnaire)
2. Non-invasive Tear Break-up Time (NIKBUT)- Oculus K5M
3. Conjunctival Redness- Oculus K5M
4. Tear collection from Schirmers strip
5. Impression Cytology- using EyePrim conjunctival membranes
6. Corneal Fluorescein Staining- Oculus K5M
7. In vivo corneal confocal microscopy (CCM)
8. Retrieval of clinical information from participants

ELIGIBILITY:
Inclusion criteria:

Recruitment inclusion criteria for Systemic diseases participants:

1. Clinically diagnosed with Primary Sjogren's Syndrome, Rheumatoid Arthritis or Systemic Lupus Erythematosus.

Recruitment inclusion criteria for controls:

1. NO Dry eye or severe Meibomian Gland Disease
2. NO current or recent (< 6 months) conjunctivitis, keratitis, uveitis or other inflammatory condition affecting eye
3. NO recent ocular surgery or LASIK (< 6 months)
4. Frequency of dry eye symptoms is < once/week (burning, tearing, itching, foreign body sensation, transient blurring improved by blinking)
5. NO contact lens wear for the past 1 week
6. NO systemic conditions of Diabetes Mellitus, Rheumatoid Arthritis, Systemic Lupus Erythematosus
7. Bulbar redness is < 1.5 grading

Exclusion Criteria:

1. Known history of thyroid disorders (diagnosed by physician)
2. No ocular surgery within the last 3 months and LASIK within 1 year.
3. Ocular surface diseases such as pterygium, or obvious lid/orbital disease with lagophthalmos.
4. Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit patients with 3 specific rheumatological diagnoses and controls
  * SS (n=40), RA (n=40), SLE (n=40)
  * Healthy age/ethnicity/sex matched control subjects (n=40)
  Total sample size: 160
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Dry Eye Symptoms (SPEED Questionnaire) | Day 0

SECONDARY OUTCOMES:
Non-invasive Tear Break-up Time (NIKBUT) | Day 0
Conjunctival Redness Grading with Oculus Keratograph 5M | Day 0
Tear collection from Schirmers strip | Day 0
To profile immune cells with EyePRIM membrane | Day 0
  Patients will be instilled with 1 drop of local anaesthetic. Conjunctival cells will be collected using EyePrim membrane by applying the membrane on the temporal and nasal conjunctival, the conjunctival cells will then be scrapped off the membrane using a 10ul micropipette tip into the 1.5ml of RPMI solution in a 2ml eppendorf tube. On the same day, FACs analysis will be done on the cells in the lab.
Documenting Corneal Fluorescein Staining | Day 0
Measuring cornea nerve density | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Cynthia Boo, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No